CLINICAL TRIAL: NCT07033949
Title: A Randomized Controlled Study on the Effect of Green Light Exposure at Different Times on the Pain of Subjects
Brief Title: Effect of Green Light Exposure at Different Times on the Pain of Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GLE
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pain
Keywords: Acute Pain; Green light
MeSH Terms: conditions — Pain; Acute Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green light exposure group (Experimental): Before performing the arterial puncture, expose to green light for 30 minutes.
  Interventions: Device: Green light glasses
- Transparent light exposure (Placebo Comparator): Before performing the arterial puncture, expose to Transparent light for 30 minutes.
  Interventions: Device: Transparent light exposure

INTERVENTIONS:
Device: Green light glasses — Exposure to green light for 30 minutes
  Arms: Green light exposure group
Device: Transparent light exposure — Exposure to transparent light for 30 minutes
  Arms: Transparent light exposure

SUMMARY:
Patients who met the criteria and needed to undergo elective surgery via arterial and venous puncture were included in this center. They were randomly divided into three time periods (8:00-9:00, 12:00-13:00, 16:00-17:00) and were exposed to green light (experimental group) and transparent light (control group) respectively. The effects of green light exposure on acute perioperative pain in patients were observed at different times.

DETAILED DESCRIPTION:
Random numbers were generated by the computer to randomly assign patients who met the inclusion and exclusion criteria to the experimental group (exposed to green light) and the control group (exposed to transparent light). The patients were randomly assigned to three time periods (8:00-9:00, 12:00-13:00, 16:00-17:00) to receive a colored exposure with glasses: Therefore, in order to minimize bias and expectations, it was not informed to the patients which color would affect the pain during the arterial puncture. The patients rested in the pre-anesthesia room for 5 minutes, their heart rate (HR) was measured, and a pain sensitivity test (tender point) was conducted. Then, the patients wore the trial glasses and stayed in the pre-anesthesia room for 30 minutes, and they underwent arterial and venous punctures. While monitoring the patients' heart rate, the catheterization of the arterial and venous punctures was performed. Then, during the arterial and venous puncture, their pain scores (NRS) were recorded separately.

exposed to green light (green group) for 30 minutes. The above operation will be repeated to measure the patient's pain threshold.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18 - 50 years old.
2. ASA classification: I - III.
3. Planned to undergo abdominal surgeries requiring general anesthesia and arterial puncture (this is not necessary for the healthy volunteer group).
4. Obtained informed consent from the patients.

Exclusion Criteria:

1. Skin ulceration, allergic reactions, or dermatitis at the tested area.
2. Long-term use of analgesics or psychiatric medications.
3. History of color blindness or uncorrected cataracts.
4. Severe cardiovascular or respiratory diseases, inflammatory disorders, etc.
5. Failure of the first arterial puncture.
6. Communication difficulties, etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during arteriovenous puncture | The pain score during arterial puncture which about 2-3min
  assessed using number rating scale (0 to 10, which higher scores mean a worse pain intensity)

SECONDARY OUTCOMES:
Pain sensitivity | from the time before to 30 min after light exposure
  assessed by pressure pain stimulation (magnitude of pressure, kilogram per square centimeter)
Analgesic consumption during surgery | From surgery beginning to the ending of the surgery
  assessed by the actual dose of analgesic during the surgery
Pain intensity after surgery | From ending of the surgery to 24 hours after surgery
  assessed using number rating scale (0 to 10, which higher scores mean a worse pain intensity)
Analgesic consumption after surgery | From ending of the surgery to 24 hours after surgery
  assessed by the actual dose of analgesic after surgery

OTHER OUTCOMES:
Heart rate | from before arterial puncture to 5min after the arterial puncture
  assessed by the monitor using beat per minute

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China